CLINICAL TRIAL: NCT00636350
Title: Bioavailability of Pepper Carotenoids in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Guangwen Tang, Tufts University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 58-1950-7-707
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2009-09

CONDITIONS: Healthy
Keywords: pepper carotenoids; xanthophylls; healthy volunteers
MeSH Terms: interventions — Lutein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Pepper — pepper carotenoids as meals
  Other Names: lutein; xanthaphylls

SUMMARY:
- list item one, Peppers

We propose to evaluate bio absorption of pepper carotenoids in a red bell-pepper or non-pungent green jalapeno pepper. The pepper will be provided in a cooked dish. The specific aims of this study are: 1) to determine blood response kinetics of lutein following multiple doses of non-pungent green jalapeno pepper with meals. 2) to determine blood response kinetics of zeaxanthin/capsanthin following multiple doses of red bell pepper with meals. We will feed 16 healthy man and women (50 - 65 y, females were at least one year post menopause), each cooked green jalapeno pepper or red pepper for 4 days and donate blood samples up to 21 days to determine blood response kinetics of xanthophylls following multiple doses of pepper dishes.

DETAILED DESCRIPTION:
- list item one, Peppers

Epidemiological data show that carotenoids and ß-C are health promoting when taken at physiologic levels in foods. However, human absorption and metabolism of carotenoids contained in various food matrices has not been studied well. It is important to investigate the characteristics of absorption and disposal kinetics after eating carotenoid rich foods in order to gain a basic understanding of the biological characteristics of lutein, zeaxanthin, and other carotenoids in food sources.

We propose to evaluate bio absorption of pepper carotenoids in a 2-phase research study: phase 1 will utilize red bell-pepper and phase 2 will utilize non-pungent green jalapeno pepper. The pepper will be provided as a dish in a meal. We will feed 16 healthy man and women (50 - 70 y, females were at least one year post menopause), each with red pepper (phase 1) and/or green jalapeno pepper (phase 2) for ~ 4 days and donate blood samples up to 21 days. Volunteers will be randomly assigned to one of the following two phases: phase 1 and phase 2.

The study will provide us the information on the bioavailability of pepper carotenoids.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* GI track problems

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-06-30 (Actual); Study Completion 2010-06-30 (Actual)

PRIMARY OUTCOMES:
The enrichment of labeled pepper carotenoids in the serum samples after the meals. | upto 21 days after the start of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts University, Boston, Massachusetts, United States